

## คณะกรรมการพิจารณาจริยธรรมการวิจัย คณะแพทยศาสตร์ จุฬาลงกรณ์มหาวิทยาลัย

## เอกสารแสดงความยินยอมเข้าร่วม โครงการสำหรับอาสาสมัคร

AF 06-07/6.1

หน้า 1/2

Research title: Effectiveness of Low Level Light Therapy and Intense Pulse Light on Mite Count as Adjuntive Therapies in Demodex Blepharitis Using Artificial Intelligent Program (Ai-Demodex): A Factorial Randomized Sham-Controlled Trial

| Date: Month: Year: |
|---|
| , Mr./Mrs./Ms, |
| residing at, |
| nave read and understood the details provided in the attached Participant Information Sheet dated |
| and voluntarily consent to participate in this research study. |

I have received a copy of the signed consent form along with the Participant Information Sheet. Prior to signing this consent form, I was provided with a thorough explanation by the researcher regarding the study's objectives, duration, research methods, potential risks or adverse effects from the study or the medication used, as well as the expected benefits of the study and alternative treatment options. I had sufficient time and opportunity to ask questions and clarify any doubts, and the researcher answered all my questions willingly and transparently until I was fully satisfied.

I have been informed by the researcher that, in the event of any harm resulting from the study, I will receive medical treatment at no cost.

I understand that I have the right to withdraw from the study at any time without providing a reason, and such withdrawal will not affect my medical treatment or any other rights I am entitled to.

The researcher assures that my personal information will be kept confidential and will only be disclosed with my consent. However, representatives from the research sponsor, the Ethics Review Committee, and the Food and Drug Administration may be permitted to access and review my data solely for the purpose of verifying the accuracy of the study. By agreeing to participate in this study, I consent to the review of my medical records for research validation purposes.

The researcher guarantees that no additional data will be collected after I withdraw from the study, and upon my request, any documents and/or samples that could identify me will be destroyed.

I understand that I have the right to review or modify my personal information and withdraw my consent for the use of my personal data at any time by notifying the researcher.

I acknowledge that my research data, including anonymized medical information, will be processed through various stages such as data collection, recording in study logs and computer systems, validation,



## คณะกรรมการพิจารณาจริยธรรมการวิจัย คณะแพทยศาสตร์ จุฬาลงกรณ์มหาวิทยาลัย

## เอกสารแสดงความยินยอมเข้าร่วม โครงการสำหรับอาสาสมัคร

AF 06-07/6.1

หน้า 2/2

analysis, and reporting for academic purposes. Furthermore, my medical and research data may be used in future studies or pharmaceutical research without requiring additional consent.

I have read and fully understood the above information and voluntarily agree to participate in this study. Therefore, I sign this consent form as confirmation of my willingness to participate.

| Signature of Participant: |
|---|
| (Printed Name:) |
| Date: Month: |
| I have explained the study's objectives, methodology, potential risks or adverse effects from the research or medication used, and the expected benefits in detail to the participant named above. The participant has acknowledged and understood the information provided and has willingly signed this consent form. |
| Signature of Researcher: |
| (Printed Name:) |
| Date: Month: |
| Signature of Witness: |
| (Printed Name: |
| Date: Month: |